CLINICAL TRIAL: NCT03757039
Title: Multifocal Visual Performance Study - Seamless Transition With Precision Profile MF Lenses
Brief Title: Multifocal Visual Performance Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLT792-P001
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Presbyopia
Keywords: contact lenses; multifocal; spectacles; glasses; progressive; vision; eyes
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This was a double-masked trial for the contact lens wearers. The PAL wearers were not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Multifocal Contact Lenses (Experimental): Multifocal soft contact lenses according to the subject's prescription and fitted using the Alcon multifocal fitting guide. Lenses were worn bilaterally (in both eyes) for up to 3 hours, 1 day only.
  Interventions: Device: Multifocal soft contact lenses
- PAL Spectacles (Active Comparator): Progressive addition lens spectacles according to the subject's habitual prescription, with testing up to 3 hours, 1 day only.
  Interventions: Other: Progressive addition lens spectacles

INTERVENTIONS:
Device: Multifocal soft contact lenses — Commercially available contact lenses
  Other Names: DAILIES TOTAL1® Multifocal contact lenses (DT1 MF); DAILIES® AquaComfort Plus® Multifocal contact lenses (DACP MF); AIR OPTIX® plus HydraGlyde® Multifocal contact lenses (AOHG MF)
  Arms: Multifocal Contact Lenses
Other: Progressive addition lens spectacles — Per subject's habitual prescription
  Other Names: PAL
  Arms: PAL Spectacles

SUMMARY:
The purpose of this trial was to compare the functional visual performance of Precision Profile Multifocal (MF) contact lenses to Progressive Addition Lens (PAL) spectacles in a presbyopic population.

DETAILED DESCRIPTION:
Habitual contact lens wearers were randomized 1:1:1 to one of three commercially available multifocal contact lenses. Progressive addition lens wearers wore their habitual spectacles. Subjects were expected to attend 1 or 2 office visits. This study was terminated early by Alcon due to slow enrollment and inconsistency in measurement of the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Normal eyes, other than correction for refractive error;
* Habitual correction of either any multifocal contact lens with a maximum add of +2.00 Diopter (D), or progressive addition lens spectacles with a maximum add of +2.00 D;
* Wears habitual correction at least 5 days per week and at least 6 hours per day.

Exclusion Criteria:

* Monocular subjects;
* Subjects fit with only one contact lens;
* Known pregnancy or lactating;
* History of or planned refractive surgery or irregular cornea in either eye.

Other protocol-specified inclusion and/or exclusion criteria may apply.

Ages: 38 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Clinical Manager, CDMA, Study Director — Alcon Research, LLC
Locations (2):
- Alcon Investigative Site, Houston, Texas, United States
- Alcon Investigative Site, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at investigative sites located in the United States (1) and United Kingdom (1).
Pre-assignment Details: Of the 42 enrolled, 1 subject was exited from the study as a screen failure prior to randomization. This reporting group includes all randomized/assigned subjects (41).
Groups:
- Multifocal Contact Lenses: All subjects randomized to multifocal contact lenses (AOHG MF, DT1 MF, or DACP MF)
- PAL Spectacles Wearers: All subjects assigned to progressive addition lens (PAL) spectacles
Period: Overall Study
Arm/Group | Multifocal Contact Lenses | PAL Spectacles Wearers
Started | 32 | 9
AOHG MF (AOHG MF = AIR OPTIX plus HydraGlyde Multifocal contact lenses) | 11 | 0
DT1 MF (DT1 MF = DAILIES TOTAL1 Multifocal contact lenses) | 11 | 0
DACP MF (DACP MF = DAILIES AquaComfort Plus Multifocal contact lenses) | 10 | 0
Completed | 32 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects exposed to any study product evaluated in this study, except for the lenses used at Visit 2 for the purpose of parameter optimization and fitting, as they are not intended for the assessment of safety (Safety Analysis Set).
Groups:
- AOHG MF: All subjects randomized to AOHG MF
- DT1 MF: All subjects randomized to DT1 MF
- DACP MF: All subjects randomized to DACP MF
- PALs: All subjects assigned to PALs
- Total: Total of all reporting groups
Arm/Group | AOHG MF | DT1 MF | DACP MF | PALs | Total
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (4.1) | 52.5 (4.1) | 51.9 (4.0) | 51.7 (3.6) | 52.0 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 6 | 5 | 24
  Male | 6 | 3 | 4 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 8 | 8 | 7 | 3 | 26
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Transition Time, Calculated From a Maximum of 3 Readings, Recorded in Seconds, During Alternate Viewing From Distance (4 m) to Intermediate (80 cm) and Vice Versa (Full Analysis Set)
Description: The subject was asked to read text at distance (4 meters) or intermediate (80 centimeters), followed immediately by text at the alternate viewing (intermediate or distance). The interval between when the subject stopped reading the first text and started reading the second text is defined as the transition time. Due to inconsistent measurement of the primary endpoint in this study, interpretation of the average transition times was compromised and the planned inferential analysis was not carried out.
Time Frame: Day 1, after up to 3 hours of wear
Population: This analysis population includes all subjects assigned to PALs or randomized to the contact lens group who were exposed to any study product evaluated in this study, except for the lenses used for optimization and fitting (Full Analysis Set).
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Multifocal Contact Lenses: Multifocal soft contact lenses (AOHG MF, DACP MF, DT1 MF combined) according to the subject's prescription and fitted using the Alcon multifocal fitting guide. Lenses were worn bilaterally (in both eyes) for up to 3 hours, 1 day only.
Arm/Group | Multifocal Contact Lenses | PAL Spectacles
Number analyzed (Participants) | 32 | 9
seconds | 2.602 (1.136) | 2.774 (0.839)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment until study exit, typically up to approximately 14 days.
Description: This analysis population includes all subjects exposed to any study product evaluated in this study, except for the lenses used at Visit 2 for the purpose of parameter optimization and fitting, as they are not intended for the assessment of safety (Safety Analysis Set).
Groups:
- AOHG MF: All subjects exposed to AOHG MF
- DT1 MF: All subjects exposed to DT1 MF
- DACP MF: All subjects exposed to DACP MF
- PALs: All subjects exposed to PALs
Arm/Group | AOHG MF | DT1 MF | DACP MF | PALs
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AOHG MF (N=11) | DT1 MF (N=11) | DACP MF (N=10) | PALs (N=9)
Blurred Vision (Eye disorders) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to inconsistent measurement of the primary endpoint in this study, interpretation of the average transition times was compromised.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT03757039/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03757039/SAP_001.pdf